CLINICAL TRIAL: NCT04761848
Title: Evaluation the Safety and Efficacy of Cilostazol in Treatment of Patients With Fatty Liver Disease: A Randomized, Controlled Trial.
Brief Title: Evaluation the Safety and Efficacy of Cilostazol in Treatment of Patients With Fatty Liver Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2021IRI
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol (Experimental)
  Interventions: Drug: Cilostazol 50 MG
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol 50 MG — Cilostazol 50 MG tablet twice daily
  Arms: Cilostazol
Drug: Placebo — Placebo tablet twice daily
  Arms: Placebo

SUMMARY:
The aim of the current study is to evaluate the safety and efficay of cilostazol in treatment of patients with fatty liver disease. Several previous reports have shown that cilostazol ameliorates lipid imbalances in NAFLD. Cilostazol appeared to exert beneficial effects against NAFLD

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 60 years of age, both men and women,
* Clinical diagnosis of NAFLD, confirmed by imaging exams,
* Patients who present levels above the reference values of ALT, AST and ferritin.

Exclusion Criteria:

* Women in the menacing period, with the exception of those who have performed definitive sterilization, such as hysterectomy or tubal ligation.
* Patients with established prior diagnosis of chronic noncommunicable disease (congestive heart failure, decompensated or severe lung disease, neoplasms, renal disease, advanced liver disease - Child Pugh C classification)
* Patients with schistosomiasis;
* Hemochromatosis
* Wilson's disease
* Viral or autoimmune hepatitis
* HIV virus carriers
* Woman who is breastfeeding
* Users of illicit drugs
* Patients with an intake of more than 20 g / day of alcohol and / or past alcoholism with abstention less than 6 months;
* Patients with ingestion of medications such as steroids, estrogens, amiodarone, warfarin, anti-convulsants, antipsychotics, tamoxifen or other chemotherapeutic agents in the last 6 months
* Patients with clinically manifest infections or inflammation, surgery, trauma or hospitalization in the last 30 days
* Chronic non-hepatic degenerative diseases (sclerosis, Parkinson's disease or -Alzheimer's disease)
* Patients who do not participate in all stages of the research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hepatic transaminases | week 12
  Alanine aminotransferase (ALT) and Aspartate Aminotransferase (AST) will be evaluated in U/L
Serum ferritin | week 12
  Serum ferritin

SECONDARY OUTCOMES:
Lipid profile | week 12
  Total cholesterol (mg/dL), LDL-cholesterol (mg/dL), HDL-cholesterol (mg/dL), VLDL-cholesterol (mg/dL) and triglycerides (mg/dL) will be measured before and after the intervention.
Glycated haemoglobin | week 12
  Hb A1c (%)
Serum stem cell transforming factor beta | 12 weeks
  Serum stem cell transforming factor beta
Adverse effects | 12 weeks
  Adverse effects
FAM19A5 serum level | 12 weeks
  FAM19A5 serum level

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF